CLINICAL TRIAL: NCT06211907
Title: Small Macular Holes Treated With Air: A Prospective Randomized Controlled Multicenter Trial
Brief Title: Small Macular Holes Treated With Air
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Haukeland University Hospital (Other); St. Olavs Hospital, Trondheim, Norway (Unknown); Oslo University Hospital, Oslo, Norway (Unknown); University Hospital of Northern Norway, Tromsø, Norway (Unknown); University of Stavanger (Other); Royal Liverpool University Hospital (Other Government); Bangor University, Qwynedd, UK (Unknown); McGill University (Other); University Hospital Complex of Santiago de Compostela, Galicia, Spain (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REK 580226
Record Dates: First submitted 2023-11-20; First posted 2024-01-18 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Macular Holes
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Intervention Model Description: Non-inferiority Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gas tamponade (Active Comparator): Intravitreal gas tamponade
  Interventions: Device: Postoperative intraocular tamponade
- Air tamponade (Experimental): Intravitreal Air tamponade
  Interventions: Device: Postoperative intraocular tamponade

INTERVENTIONS:
Device: Postoperative intraocular tamponade — Flushing the eye cavity with a tamponade at the end of surgery

SUMMARY:
Non-inferiority trial comparing intraocular air and gas tamponade for closure of macular holes.

ELIGIBILITY:
Inclusion Criteria:

* Primary MH ≤250 μm
* MH duration ≤12 months
* No previous vitreoretinal surgery in study eye
* Ability to sign informed consent
* Signed informed consent
* Age ˃18 years

Exclusion Criteria:

* Previous vitreoretinal surgery in study eye
* Secondary MH caused by other conditions than vitreomacular traction
* Myopic MH, i.e., excessive myopia (more than -6 dioptres)
* Traumatic MH
* MH secondary to retinal detachment or other retinal diseases
* Previously participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-07-14 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Macular hole closure after single surgery | 4 weeks
  Closure verified on OCT

SECONDARY OUTCOMES:
Change in outcome of patient well-being | 4 weeks and 4 months
  Questionnaire
Change in visual acuity i ETDRS lines | 4 weeks and 4 months
  Early Treatment of Diabetic Retinopathy Score in logMAR. Higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Locations (7):
- Department of Ophthalmology, University of Thessaly, Thessaly, Thessaly, Greece
- Norway (5):
  - Stavanger University Hospital, Stavanger, Rogaland
  - University Hospital of Northern Norway, Tromsø, Troms
  - St. Olavs University Hospital, Trondheim, Tronderlag
  - Haukeland University Hospital, Bergen, Vestland
  - Oslo University Hospital, Oslo
- Clinical Universitary Hospital of Santiago, Santiago de Compostela, La Coruna, Spain